CLINICAL TRIAL: NCT02204085
Title: A Phase I/II Trial of the MUC1 Inhibitor, GO-203-2C in Patients With Relapsed or Refractory Acute Myeloid Leukemia
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Beth Israel Deaconess Medical Center (Other)
Collaborators: Dana-Farber Cancer Institute (Other)
Responsible Party: Principal Investigator, David Avigan, Principal Investigator, Beth Israel Deaconess Medical Center
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 14-222
Record Dates: First submitted 2014-07-09; First posted 2014-07-30 (Estimated); Last update posted 2025-01-24 (Actual); Status verified 2025-01

CONDITIONS: Acute Myeloid Leukemia, in Relapse; Recurrent Adult Acute Myeloid Leukemia
Keywords: Refractory acute myeloid leukemia; Relapsed acute myeloid leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — Decitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- GO-203-2c (Experimental): Dose escalation will occur using a standard 3+3 dose escalation approach, beginning in dose level I with dose cohorts and rules for escalation and de-escalation.
  GO-203-2c given daily on predetermined schedule of a 28-day treatment cycle
  Interventions: Drug: GO-203-2c
- GO-203-2c + Decitabine (Experimental): Dose escalation will occur for GO-203-2c using a standard 3+3 dose escalation approach, beginning in dose level I with dose cohorts and rules for escalation and de-escalation.
  GO-203-2c given daily on predetermined schedule of a 28-day treatment cycle. Decitabine will be administered at a dose of 20mg/m2 on days 8-12 of a 28-day treatment cycle.
  Interventions: Drug: GO-203-2c; Drug: GO-203-2c + Decitabine

INTERVENTIONS:
Drug: GO-203-2c
Drug: GO-203-2c + Decitabine
  Arms: GO-203-2c + Decitabine

SUMMARY:
This research study is studying a targeted therapy known as GO-203-2C as a possible treatment for with acute myeloid leukemia (AML) both alone and in combination with decitabine. GO-203-2c targets cancer cells, while leaving healthy cells unaffected.This is a Phase I/II clinical trial. A Phase I clinical trial tests the safety of an investigational intervention and also tries to define the appropriate dose of the investigational intervention to use for further studies.

DETAILED DESCRIPTION:
* Phase I

  * The maximum tolerated dose (MTD) will be determined in the phase I section of the trial.
  * Patients who fulfill eligibility criteria will be entered into the trial to GO-203-2c.
  * After the screening procedures confirm participation in the research study. The investigators are looking for the highest dose of the combination of study drugs that can be administered safely without severe or unmanageable side effects in participants that have acute myeloid leukemia (AML) not everyone who participates in this research study will receive the same dose of the study drug. The dose given will depend on the number of participants who have been enrolled in the study prior and how well the dose was tolerated.
  * A subsequent dose escalation will evaluate the combination of GO-203-2c and decitabine.
* Phase II

  * The primary goal is to determine if the combination of the two drugs results in clinical response

ELIGIBILITY:
Inclusion Criteria:

* To be considered eligible for enrollment into this study, all of the following inclusion criteria must be met during the screening period:
* Documented AML by peripheral blood and bone marrow analyses meeting WHO criteria, excluding patients with acute promyelocytic leukemia (APL)
* Patients with AML refractory to primary induction chemotherapy, relapsed disease, or age ≥ 60 and not appropriate for standard cytotoxic therapy due to age, performance status, and/or adverse risk factors according to the treating physician
* Age ≥ 18 years
* Karnofsky performance status ≥ 50% or ECOG performance status 0-2
* Life expectancy ≥ 6 weeks
* Able to understand the investigational nature of this study and to provide written consent to participate in it
* Signed written IRB-approved Informed Consent document
* Adequate hepatic and renal function:

  * serum bilirubin ≤ 1.5 X institutional ULN OR serum direct bilirubin ≤ 2 X institutional ULN
  * serum ALT and AST ≤ 2.5 X institutional ULN
  * serum alkaline phosphatase < 5 X institutional ULN
  * serum creatinine ≤ 2.0 mg/dL
  * corrected calcium level ≥ institutional LLN
* Negative pregnancy test in women of child-bearing potential
* Women and men of child-producing potential must agree to use effective contraceptive methods during the study period (including post-treatment observation period)

Exclusion Criteria:

* A patient will be considered not eligible for enrollment into this study if any of the following criteria are met during the screening period:
* Evidence of leukemic meningitis or other CNS involvement by leukemia
* Uncontrolled or poorly controlled hypertension (systolic BP ≥ 160 mmHg or diastolic BP ≥ 100 mmHg) Note: an isolated reading that is not sustained will be permitted.
* Evidence of NYHA Class III or IV cardiac disease, or presence of unstable life-threatening arrhythmia, or history of myocardial infarction during the past 6 months
* Active bacterial, fungal, or viral infection requiring systemic treatment
* Known infection with HIV
* History or major surgery within 4 weeks before the first dose of study treatment, or not recovered from prior surgery
* Exposure to any other investigational agent at any time within 4 weeks before the first dose of study treatment
* Exposure to any other anti-leukemic therapy (except hydroxyurea, see Section 5.5.1) within 2 weeks before the first dose of study treatment
* Pregnant or lactating female
* Unwilling or unable to comply with the requirements of the study protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2014-09; Primary Completion 2025-09 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Maximum Tolerated Dose of GO-203-2c | 28 days
  Phase I
Maximum Tolerated Dose of GO-203-2c in combination with decitabine | 28 days
  Phase 1

SECONDARY OUTCOMES:
Number of Participants with Adverse Events as a Measure of Safety and Tolerability | 2 years
To investigate whether GO-203-2c alone and in combination with decitabine is effective in targeting MUC1-C overexpressing AML progenitor cells in the lab | 2 Years
To assess whether in vitro response to GO-203-2c alone and in combination with decitabine is associated with clinical response | 2 Years
To determine if therapy with GO-203-2c alone and in combination with decitabine results in decreased engraftment potential of AML progenitor cells in an NSG mouse model | 2 Years
To determine if therapy GO-203-2c in combination with decitabine results in at least 20% of patients achieving a clinical response | 2 years
  To determine if therapy GO-203-2c in combination with decitabine results in at least 20% of patients achieving a clinical response (blast response, minor response, partial response, or complete response).

CONTACTS AND LOCATIONS:
Overall Officials: David Avigan, MD, Principal Investigator — Beth Israel Deaconess Medical Center
Locations (2):
- United States (2):
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts